CLINICAL TRIAL: NCT00646373
Title: Effect of Decreased Pump Prime Volume on Blood Transfusions and Postoperative Complications of Patients Undergoing High Risk Cardiac Surgical Procedures: A Pilot Study
Brief Title: Effect of Decreased Pump Prime Volume on Blood Transfusions and Postoperative Complications of Patients Undergoing High Risk Cardiac Surgical Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol was comparing to standard of practice, which has changed over the course of slow recruitment and no longer can be used as a comparator.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Massimiliano Meineri, Toronto General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHN REB#06-0012-B
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2006-12

CONDITIONS: Cardiac Surgery
Keywords: Cardiac surgery; Pump prime; Blood transfusions

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Other: Low Prime — The CPB circuit will be primed with mannitol (50 g of 20% solution) and crystalloid solution (Ringer's lactate) for a total volume of approximately 1200 ml.

SUMMARY:
The objective of this study is to evaluate the impact of reduced pump prime on blood transfusions and postoperative complications in patients at high risk of severe hemodilution during CPB.

HYPOTHESIS The use of a new CPB circuit with a smaller internal volume, together with retrograde autologous priming of the lines (RAP) will allow a smaller prime volume and therefore less significant hemodilution on pump.

EXPERIMENTAL DESIGN Overview

Patients will be randomized on the morning of surgery to one of the two study groups in a 1:1 allocation scheme:

1. Low pump prime
2. Standard pump prime Outcomes The primary outcome is the number of units of blood products transfused within the first 24 hours post CPB.

ELIGIBILITY:
Inclusion Criteria:

* >18 y of age
* Non-emergent complex cardiac surgery (any procedure other than primary isolated CABG)
* Any of the following: Hb < 120 g/L (Females) or < 130 g/L (Males)BSA < 1.6 m2Creatinine Clearance < 60 mL/min (Cockcroft Gault Equation)

Exclusion Criteria:

* aPTT >50 s, INR>1.5
* Plt < 100,000 x 106
* Preoperative Hemodialysis
* Tight aortic stenosis (Aortic Valve Area < 1 cm2)
* Tight lesion of the left main coronary artery (> 60%)
* Use of Aprotinin requested by the Surgical Team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The number of units of blood products transfused within the first 24 hours post CPB. | 24 hours